CLINICAL TRIAL: NCT01556542
Title: Drug Eluting Balloon in peripherAl inTErvention: the DEBATE SFA Study
Brief Title: Drug Eluting Balloon in peripherAl inTErvention SFA
Acronym: DEBATE SFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leonardo Bolognese, MD (Other)
Responsible Party: Sponsor-Investigator, Leonardo Bolognese, MD, Director of Cardiovascular Department, Ospedale San Donato
Organization: Ospedale San Donato (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arezzo004
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; drug-eluting balloon; restenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard PTA (Active Comparator): nitinol stent implantation
  Interventions: Device: nitinol stent implantation
- DEB (Experimental): paclitaxel-eluting balloon angioplasty followed by nitinol stent implantation
  Interventions: Device: paclitaxel-eluting balloon angioplasty followed by nitinol stent implantation

INTERVENTIONS:
Device: paclitaxel-eluting balloon angioplasty followed by nitinol stent implantation — paclitaxel-eluting balloon angioplasty followed by nitinol stent implantation
  Arms: DEB
Device: nitinol stent implantation — nitinol stent implantation
  Arms: standard PTA

SUMMARY:
The purpose of this study is to evaluate the efficacy of drug-eluting balloon angioplasty followed by nitinol stent implantation versus nitinol stent implantation in superficial femoral artery and popliteal artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* intermittent claudication(Fontane III or IV)
* angiographic stenosis>50% or occlusion of superficial femoral-popliteal artery>40mm
* at least one below-knee vessel to the ankle

Exclusion Criteria:

* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
angiographic binary restenosis | 12 months
  incidence of binary restenosis

SECONDARY OUTCOMES:
major amputation | 24 months
  incidence of major amputation
target lesion revascularization | 24 months
  incidence of target lesion revascularization
vessel reocclusion | 24 months
  incidence of vessel reocclusion

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Liistro, MD, Principal Investigator — Cardiovascular Department, San Donato Hospital, Arezzo, Italy
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Liistro F, Grotti S, Porto I, Angioli P, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for the superficial femoral artery: the DEBATE-SFA randomized trial (drug eluting balloon in peripheral intervention for the superficial femoral artery). JACC Cardiovasc Interv. 2013 Dec;6(12):1295-302. doi: 10.1016/j.jcin.2013.07.010. Epub 2013 Nov 13. PMID 24239203